CLINICAL TRIAL: NCT01189890
Title: A Phase III, Multicenter, Double-Blind, Randomized, Active-Controlled Study to Evaluate the Safety and Efficacy of Sitagliptin Compared With Glimepiride in Elderly Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control
Brief Title: Safety and Efficacy of Sitagliptin Compared With Glimepiride in Elderly Participants With Type 2 Diabetes Mellitus (MK-0431-251)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-251
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, Hemoglobin A1C, glucagon-like peptide 1 (GLP-1), gastric inhibitory polypeptide (GIP), dipeptidyl peptidase 4 inhibitor (DPP-4)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin phosphate 100 mg or 50 mg once daily (QD)
  Interventions: Drug: sitagliptin phosphate; Drug: Placebo to Glimepiride
- Glimepiride (Active Comparator): Glimepiride 1-6 mg QD
  Interventions: Drug: Glimepiride; Drug: Placebo to Sitagliptin

INTERVENTIONS:
Drug: sitagliptin phosphate — Sitagliptin tablets, orally, at a dose of 100 mg or 50 mg QD for 30 weeks. The dose level to be administered will depend on the participant's estimated glomerular filtration rate (eGFR), calculated at Visit 3 and may be adjusted as medically indicated during the study.
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Glimepiride — Glimepiride tablets, orally, starting at a dose of 1 mg QD, which may be gradually increased, as needed, to maximum dose of 6 mg QD for 30 weeks. The dose may also be decreased as medically indicated during the study.
  Other Names: Amaryl
  Arms: Glimepiride
Drug: Placebo to Sitagliptin — Matching placebo tablets to sitagliptin to allow for blinding.
  Arms: Glimepiride
Drug: Placebo to Glimepiride — Matching placebo tablets to glimepiride to allow for blinding.
  Arms: Sitagliptin

SUMMARY:
The primary objectives of this study are to determine if sitagliptin treatment is not inferior to that of glimepiride as measured by the change in baseline hemoglobin A1C (HbA1C) after 30 weeks of treatment, and if sitagliptin treatment results in a lower incidence of symptomatic hypoglycemia compared to that of glimepiride. The study will also evaluate if sitagliptin treatment, compared to glimepiride results in improvements in fasting plasma glucose (FPG) levels, and plasma lipid levels after 30 weeks of treatment. Participants will be randomized to either sitagliptin or glimepiride treatment after eligibility for study participation is determined during screening and washout study phases. Participants and study staff will not know to which treatment group they have been randomized (double-blind design). The duration of study participation will be up to 40 weeks (with 9 clinic visits). This will include a screening phase (Visit 1 to Visit 2) of 2 weeks maximum; a 6-week (Visits 2 to 3) oral antihyperglycemic agent (AHA) wash-out phase (for those who have been taking a AHA prior to the study); a placebo run-in phase (Visits 3 to 4), followed by up to 30 weeks of treatment with study medication.

DETAILED DESCRIPTION:
The dose of sitagliptin will be 100 mg once daily (QD) or 50 mg QD based on the participant's estimated glomerular filtration rate (eGFR). The starting dose of glimepiride (1 mg QD) may be up-titrated as needed to optimize glycemic control over the first 18 weeks to a maximum dose of 6 mg/day, after which the dose will not be increased for the rest of the study (down-titration to avoid or control hypoglycemia is allowed).

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of type 2 diabetes mellitus

Exclusion Criteria

* History of type 1 diabetes mellitus
* Has undergone a surgical procedure within the prior 4 weeks.
* Current participation in, or has participated, in another study with an investigational device or compound, with the prior 12 weeks, and/or is not willing to refrain from participating in any other study while participating in this study
* Hypersensitivity or contraindication to any sulfonylurea (e.g., glimepiride) medication
* Has been on an investigational or approved dipeptidyl peptidase-4 (DPP-4) inhibitor agent (e.g., sitagliptin, saxagliptin)
* Presence of human immunodeficiency virus (HIV)
* Current participation in a weight loss program or is receiving weight loss medication
* History of blood disorder, certain cancers, heart, liver or kidney disease
* Current or past use of recreational or illicit drugs, or a history of drug abuse or dependence, or increased alcohol consumption

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 480 (Actual)
Dates: Start 2010-08-16 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-10-31 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hartley P, Shentu Y, Betz-Schiff P, Golm GT, Sisk CM, Engel SS, Shankar RR. Efficacy and Tolerability of Sitagliptin Compared with Glimepiride in Elderly Patients with Type 2 Diabetes Mellitus and Inadequate Glycemic Control: A Randomized, Double-Blind, Non-Inferiority Trial. Drugs Aging. 2015 Jun;32(6):469-76. doi: 10.1007/s40266-015-0271-z. PMID 26041585

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin: Sitagliptin phosphate 100 mg once daily (QD) or 50 mg QD
Period: Overall Study
Arm/Group | Sitagliptin | Glimepiride
Started | 241 | 239 (3 randomized glimepiride participants did not receive study drug.)
Completed | 204 | 200
Not Completed | 37 | 39
Not completed — Adverse Event | 3 | 4
Not completed — Lack of Efficacy | 7 | 2
Not completed — Lost to Follow-up | 1 | 7
Not completed — Protocol Violation | 1 | 5
Not completed — Withdrawal by Subject | 15 | 11
Not completed — Non Compliance | 0 | 1
Not completed — Physician Decision | 5 | 4
Not completed — Hyperglycemia Discontinuation Criteria | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Glimepiride | Total
Number analyzed (Participants) | 241 | 239 | 480
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (4.8) | 70.8 (4.9) | 70.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 148 | 278
  Male | 111 | 91 | 202
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — The population included all randomized participants who had a baseline HbA1c, did not take prohibited concomitant medications, had compliance >85%, and did not receive any incorrect study medication. Sitagliptin (n=197) and glimepiride (n=191).
  Percentage of HbA1c | 7.78 (0.70) | 7.78 (0.67) | 7.78 (0.69)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — The population included all randomized participants who had a baseline FPG, did not take prohibited concomitant medications, had compliance >85%, and did not receive any incorrect study medication. Sitagliptin (n=194) and glimepiride (n=191).
  mg/dL | 168.4 (31.2) | 169.7 (35.5) | 169.0 (33.3)
Body Weight [Mean (Standard Deviation); unit: kg] — All randomized participants who received at least one dose of study treatment and had a body weight measurement at baseline. Sitagliptin (n=205) and glimepiride (n=203).
  kg | 76.9 (15.1) | 75.4 (16.4) | 76.0 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Least Squares (LS) Mean Change From Baseline in Hemoglobin A1c (HbA1c) at Week 30
Description: Participant whole blood samples were collected at baseline and Week 30 to determine the LS mean HbA1c change from baseline. HbA1c is a measure of the percentage of glycated hemoglobin in the blood and provides an indication of participant blood glucose control in the 2 to 3 months prior to the evaluation.
Time Frame: Baseline and Week 30
Population: The population included all randomized participants who had a baseline HbA1c, had a HbA1c at Week 30, did not take prohibited concomitant medications, had compliance >85%, and did not receive any incorrect study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of HbA1c
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 197 | 191
Percentage of HbA1c | -0.32 (0.78) [-0.51 to -0.14] | -0.51 (0.89) [-0.69 to -0.33]
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Non-Inferiority or Equivalence — The predefined non-inferiority margin was 0.4%; ANCOVA; Controlled for treatment, estimated glomerular filtration rate (eGFR) stratum, age stratum, and baseline HbA1C; Difference in LS Means = 0.19, 95% CI 2-sided [0.03 to 0.34]

2. Primary Outcome: Number of Participants With an Adverse Event of Symptomatic Hypoglycemia Up to Week 30
Description: Symptomatic hypoglycemia was defined as an episode with clinical symptoms attributed to hypoglycemia, without regard to glucose level. Participants were instructed to complete the Hypoglycemia Assessment Log (HAL) for any symptomatic episodes he or she believed represent hypoglycemia. If a fingerstick glucose was obtained before or shortly (i.e., within a few minutes) after treating, the value was recorded in the HAL. In addition, participants were instructed to record in the HAL any fingerstick glucose values ≤70 mg/dL (≤3.9 mmol/L) regardless of the presence of clinical symptoms.
Time Frame: Up to Week 30
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 241 | 236
Participants | 2 | 11
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; p = 0.009, Miettinen & Nurminen; Stratified by estimated glomerular filtration rate (eGFR) stratum and age stratum; Difference in Percent Incidence = -3.9, 95% CI 2-sided [-7.5 to -1.2]

3. Primary Outcome: Number of Participants Experiencing An Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the
  study treatment, whether or not considered related to the use of the treatment administered.
Time Frame: Up to Week 30
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 241 | 236
Participants | 118 | 115

4. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to An AE
Description: as for outcome 3
Time Frame: Up to Week 30
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 241 | 236
Participants | 3 | 4

5. Secondary Outcome: LS Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 30
Description: Plasma samples were collected from participants after an overnight fast at baseline and Week 30 to determine the mean change from baseline in participant FPG.
Time Frame: Baseline and Week 30
Population: The population included all randomized participants who had a FPG value at baseline and Week 30, did not take prohibited concomitant medications, had compliance >85%, and did not receive any incorrect study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 194 | 191
mg/dL | -14.5 (39.0) [-21.6 to -7.4] | -21.2 (39.1) [-28.3 to -14.0]
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; ANCOVA; Controlled for treatment, eGFR stratum, age stratum, and baseline FPG; Difference in LS Means = 6.7, 95% CI 2-sided [0.7 to 12.7]

6. Secondary Outcome: Percentage of Participants With HbA1c <7.0% at Week 30
Description: Participant whole blood samples were collected at Week 30 to determine the number of participants achieving HbA1c <7.0% at Week 30. HbA1c is a measure of the percentage of glycated hemoglobin in the blood and provides an indication of participant blood glucose control in the 2 to 3 months prior to the evaluation.
Time Frame: Week 30
Population: The population included all randomized participants who had HbA1c at baseline and Week 30, did not take prohibited concomitant medications, had compliance >85%, and did not receive any incorrect study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 197 | 191
Percentage of Participants | 33.5 | 46.6
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; Miettinen & Nurminen; Stratified by eGFR stratum and age stratum; Relative Risk = 0.7, 95% CI 2-sided [0.6 to 0.9]

7. Secondary Outcome: Percentage of Participants With HbA1c <6.5% at Week 30
Description: Participant whole blood samples were collected at Week 30 to determine the number of participants achieving HbA1c <6.5% at Week 30. Hemoglobin A1c is a measure of the percentage of glycated hemoglobin in the blood and provides an indication of participant blood glucose control in the 2 to 3 months prior to the evaluation.
Time Frame: Week 30
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 197 | 191
Percentage of Participants | 9.1 | 20.9
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; Miettinen & Nurminen; Stratified by eGFR stratum and age stratum; Relative Risk = 0.4, 95% CI 2-sided [0.3 to 0.7]

8. Secondary Outcome: LS Mean Change From Baseline in Participant Body Weight at Week 30
Description: Participants were only permitted to wear a drape gown and undergarments (no street clothes, no shoes or socks) for this evaluation. Body weight was measured after voiding (to the nearest 0.1 kg) and measurements were collected until 2 consecutive measurements did not differ by more than 0.2 kg from each other. Body weight measurements were evaluated using a standardized, calibrated digital scale and was reported in kilograms (kg) at baseline and Week 30.
Time Frame: Baseline and Week 30
Population: All randomized participants who received at least one dose of study treatment and had body weight measurements at baseline and at Week 30.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 205 | 203
kg | 0.4 (3.2) [-0.2 to 1.0] | 1.1 (2.8) [0.5 to 1.7]
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; p = 0.011, ANCOVA; Controlled for treatment, eGFR stratum, age stratum, and baseline body weight; Difference in LS Means = -0.7, 95% CI 2-sided [-1.3 to -0.2]

ADVERSE EVENTS:
Time Frame: Up to Week 32.
Description: The safety population consisted of all randomized participants who received at least one dose of study treatment.
Arm/Group | Sitagliptin | Glimepiride
Serious Adverse Events (participants affected / at risk) | 7/241 | 6/236
Other Adverse Events (participants affected / at risk) | 34/241 | 40/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=241) | Glimepiride (N=236)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Chronic (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nerve Compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=241) | Glimepiride (N=236)
Nasopharyngitis (Infections and infestations) | 18 (20) | 19 (21)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (17) | 9 (15)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 15 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish results for his/her study site after publication of results of entire multicenter trial, or after public disclosure of the results online if a multicenter manuscript is not planned. Sponsor must be able to review all proposed results communications regarding study 60 days prior to submission for publication/presentation. Information identified by the Sponsor as confidential must be deleted prior to submission.